CLINICAL TRIAL: NCT02377206
Title: Neuroinflammation and Cognitive Decline in Alzheimer Disease (AD) : Pilot Study of Translocator Proteins Ligand PET Imaging With [18F]DPA-714
Brief Title: Neuroinflammation and Cognitive Decline in Alzheimer Disease
Acronym: NICAD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRTS13-CH / NICAD
Record Dates: First submitted 2015-02-17; First posted 2015-03-03 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Alzheimer Disease
Keywords: PET; [18F]DPA-714; cognitive decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alzheimer Disease (Experimental): Alzheimer Disease People ADAS-Cog evaluation PET imaging with [18F]DPA-714
  Interventions: Other: ADAS-Cog evaluation

INTERVENTIONS:
Other: ADAS-Cog evaluation — [18F]DPA-714 PET imaging

SUMMARY:
The purpose of this study is to assess the level of neuroinflammation in Alzheimer Disease subject (mild to moderate) estimated with Binding Potential (BP) of [18F]DPA-714, and its relationship with the kinetics of cognitive decline over a 24-month follow-up period (as assessed by Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) and Mini-Mental State Examination (MMSE) scores).

DETAILED DESCRIPTION:
The purpose of this study is to assess the level of neuroinflammation in Alzheimer Disease subject (mild to moderate) estimated with Binding Potential (BP) of [18F]DPA-714 , and its relationship with the kinetics of cognitive decline over a 24-month follow-up period (as assessed by ADAS-Cog and MMSE scores).

(DPA-714 : N,N-diethyl-2-[4-(2-fluoroethoxy)phenyl]-5,7-dimethylpyrazolo[1,5-a]pyrimidine-3-acetamide)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age more than 50 years (included)
* necessary knowledge of French (write and oral) to do neuropsychological tests
* Study level upper (or equal) than 7 years (considering first year of grammar-school as start)
* People with Alzheimer Disease defined as National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and the Alzheimer's Disease and Related Disorders Association (ADRDA) standards : Light to mild AD defined by Mini-Mental State Examination (MMSE) score between 15 and 25 (included)
* Social security affiliation.

Exclusion Criteria:

* MMSE score lower than 15 and upper or equal to 26
* Evolutive disease which could possibly had consequences on central nervous system
* Inflammatory disease or evolutive neoplasia and/or C reactive protein (CRP) upper than 10mg/L
* Chronic use of alchohol and/or drug
* Serious depression defined by Montgomery Asberg Depression Rating Scale (MADRS) score higher than 18
* Surgical or medical condition in the last 3 months
* Long term treatment which could possibly interfere with inflammatory process (especially the month before PET [18F]DPA-714 imaging).
* Treatment by N-Methyl-D-Aspartate antagonist
* Treatment by Minocycline
* Treatment by benzodiazepine (especially the month before PET [18F]DPA-714 imaging) (Zolpidem, zopiclone and loprazolam excepted)
* Anomaly at neurological examination which is not a classical symptom
* Contraindication to magnetic resonance imaging (RMI)
* Florbetapir[18F] hypersensibility
* Participation to an other experimental protocol with drug.
* people under guardianship

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Compare the neuroinflammation measured by fixing and layout of [18F]DPA-714 between 3 groups of patients : subjects suffering from Alzheimer disease light to mild stage, amnesiac MCI and patients suffering from isolated cognitive complaint | inclusion and 24 months

SECONDARY OUTCOMES:
Relationship passessment between [18F]DPA-714 fixing | Inclusion and 34 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent CAMUS, PhD, Principal Investigator — University Hospital of Tours
Locations (3):
- France (3):
  - university hospital of Nantes, Nantes
  - University Hospital of Rennes, Rennes
  - University Hospital of Tours, Tours

REFERENCES:
- [Background] Schmidt C, Wolff M, Weitz M, Bartlau T, Korth C, Zerr I. Rapidly progressive Alzheimer disease. Arch Neurol. 2011 Sep;68(9):1124-30. doi: 10.1001/archneurol.2011.189. PMID 21911694
- [Background] Soto ME, Andrieu S, Arbus C, Ceccaldi M, Couratier P, Dantoine T, Dartigues JF, Gillette-Guyonnet S, Nourhashemi F, Ousset PJ, Poncet M, Portet F, Touchon J, Vellas B. Rapid cognitive decline in Alzheimer's disease. Consensus paper. J Nutr Health Aging. 2008 Dec;12(10):703-13. doi: 10.1007/BF03028618. PMID 19043645
- [Background] Helmer C, Andrieu S, Peres K, Orgogozo JM, Vellas B, Dartigues JF; REAL.fr Group. Predictive value of 6-month decline in ADAS-cog for survival without severe Alzheimer's disease. Dement Geriatr Cogn Disord. 2007;23(3):168-74. doi: 10.1159/000098516. Epub 2007 Jan 11. PMID 17215578
- [Background] Lo RY, Jagust WJ; Alzheimer's Disease Neuroimaging Initiative. Vascular burden and Alzheimer disease pathologic progression. Neurology. 2012 Sep 25;79(13):1349-55. doi: 10.1212/WNL.0b013e31826c1b9d. Epub 2012 Sep 12. PMID 22972646